CLINICAL TRIAL: NCT02246855
Title: A Comparison of the Pharmacokinetics, Safety and Tolerance of Two Formulations of a Liquid IVIg (Vigam® Liquid and Gammaplex®) Using Standard and Accelerated Infusion Rates in Healthy Adult Volunteers (Three Treatment Arms)
Brief Title: A Comparison of the Pharmacokinetics, Safety and Tolerance of Two Formulations of a Liquid IVIg in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: GMX03
Record Dates: First submitted 2014-09-02; First posted 2014-09-23 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Subjects
MeSH Terms: interventions — gamma-Globulins

ARMS (3):
- Vigam® Liquid infused at up to 3mL/min (Experimental): Gammaplex® (Human Normal Immunoglobulin)
  Interventions: Biological: Gammaplex® (Human Normal Immunoglobulin)
- Gammaplex® infused at up to 3mL/min (Experimental): Gammaplex® (Human Normal Immunoglobulin)
  Interventions: Biological: Gammaplex® (Human Normal Immunoglobulin)
- Gammaplex® infused at up to 6mL/min (Experimental): Gammaplex® (Human Normal Immunoglobulin)
  Interventions: Biological: Gammaplex® (Human Normal Immunoglobulin)

INTERVENTIONS:
Biological: Gammaplex® (Human Normal Immunoglobulin)

SUMMARY:
The main object of the study is to compare the AUC0-84, of a single intravenous infusion of Vigam® Liquid (infused at the licensed rate of up to 3mL/min) with Gammaplex® (infused at up to 3mL/min and up to 6mL/min).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, normotensive, non-smoking male and female volunteers aged 18 to 60 who gave written informed consent and fulfilled all of the inclusion criteria and none of the exclusion criteria.
* Female volunteers of childbearing potential had a negative pregnancy test before entering the study and had to use either a double barrier method of contraception or use the oral contraceptive pill.
* Postmenopausal or surgically sterile female volunteers could be enrolled.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-08; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
PK parameters for serum immunoglobulin G (IgG) | Screening, pre-dose (Day 1), 15 min, 4 hr, 24 hr, 30 hr, 48 hr, Days 4, 8, 11, 15, 18, 22, 29, 36, 43, 50, 57, 71, 85

CONTACTS AND LOCATIONS:
Overall Officials: David Wessels, MBChB MBA, Principal Investigator
Locations (1):
- Clinical Pharmacology Research Unit (CPRU), Level 7, Northwick Park Hospital, Watford Road, Harrow, United Kingdom